CLINICAL TRIAL: NCT06756789
Title: Randomized Controlled Trial on Conventional Vs Tailored Limb Lengths in Laparoscopic Roux-en Y Gastric Bypass Surgery
Brief Title: Conventional Vs Tailored Limb Lengths in Laparoscopic Roux-en Y Gastric Bypass Surgery
Acronym: TAILO-R-YGB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GEM Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GemBariatricRYGB
Record Dates: First submitted 2024-06-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Metabolic Disease; Bariatric Surgery Candidate; Metabolic Surgery; RYGB
Keywords: Obesity; RYGB; Bariatric surgery; Metabolic surgery; Metabolic syndrome
MeSH Terms: conditions — Obesity; Metabolic Diseases; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional group (Placebo Comparator): In this arm, standard limb lengths of 75cms BP limb and 125cms Alimentary limb were measured and performed, irrespective of the total bowel length
  Interventions: Procedure: Laparoscopic Roux-en Y Gastric bypass (RYGB)- Conventional approach
- Tailored group (Active Comparator): In this arm, limb lengths are tailored according to the total small bowel length, 1/3rd of the total bowel length is measured and in that 3/8th and 5/8th were kept as BP limb and alimentary limb respectively.
  Interventions: Procedure: Laparoscopic Roux-en Y Gastric bypass (RYGB)- Tailored approach

INTERVENTIONS:
Procedure: Laparoscopic Roux-en Y Gastric bypass (RYGB)- Conventional approach — The procedure involves creating a small gastric pouch from the upper portion of the stomach, which is then directly connected to the small bowel, in a roux- enY fashion with another jejune-jejunal anastamosis bypassing a large part of the stomach and the duodenum. This results in reduced food intake and decreased nutrient absorption. In this arm, standard limb lengths of 75cms BP limb and 125cms Alimentary limb were measured and performed, irrespective of the total bowel length
  Arms: Conventional group
Procedure: Laparoscopic Roux-en Y Gastric bypass (RYGB)- Tailored approach — The procedure involves creating a small gastric pouch from the upper portion of the stomach, which is then directly connected to the small bowel, in a roux- enY fashion with another jejune-jejunal anastamosis bypassing a large part of the stomach and the duodenum. This results in reduced food intake and decreased nutrient absorption. In this arm, limb lengths are tailored according to the total small bowel length, 1/3rd of the total bowel length is measured and in that 3/8th and 5/8th were kept as BP limb and alimentary limb respectively.
  Arms: Tailored group

SUMMARY:
The study aims to investigate whether tailoring limb lengths based on the 1/3rd and 2/3rd concept improves clinical outcomes in Laparoscopic Roux-en-Y Gastric Bypass (LRYGB) surgery compared to conventional limb lengths. In this study, two groups were described, first group involves patients who will undergo Lap RYGB with conventional limb lengths of 75cms and 125cms, while the second group is given tailored limb lengths according to the total small bowel length. In the follow up period, Total percentage weight loss, improvement in BMI along with the remission of co-morbidities were also assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years
2. Body Mass Index (BMI):

   BMI ≥ 40 kg/m² or BMI ≥ 35 kg/m² with at least one obesity-related comorbidity (e.g., type 2 diabetes, hypertension, obstructive sleep apnea).
3. ASA - less than or equal to 3
4. Informed Consent: Ability and willingness to provide written informed consent and comply with procedures.
5. Previous Weight Loss Attempts: Documentation of previous attempts at weight loss through diet, exercise, or medical management.

Exclusion Criteria:

1. Previous Bariatric Surgery: Prior bariatric or major gastrointestinal surgery that might affect the outcome of RYGB.
2. Severe Cardiopulmonary Conditions: Significant cardiac or pulmonary conditions that pose a high surgical risk (e.g., severe congestive heart failure, severe chronic obstructive pulmonary disease).
3. Uncontrolled Psychiatric Disorders: Severe psychiatric illness or substance abuse issues that are not well-controlled, including eating disorders.
4. Pregnancy: Current pregnancy or plans to become pregnant within 12 months post-surgery.
5. Malignancy: Active malignancy or history of malignancy requiring treatment in the past 5 years (excluding non-melanoma skin cancer).
6. Severe Liver Disease: Cirrhosis or significant liver dysfunction (e.g., Child-Pugh B or C).
7. Inability to Comply: Patients who are unable or unwilling to comply with the postoperative follow-up schedule and dietary requirements.
8. Chronic Use of Medications: Chronic use of medications known to affect weight or metabolism significantly, such as corticosteroids or antipsychotics.
9. Other Medical Conditions: Any other medical condition or surgical finding that, in the opinion of the investigators, would make the patient unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of total weight loss (%TWL) | 3, 6 and 12 months
Improvement in BMI | 3, 6 and 12 months
  BMI is calculated by dividing Weight in kilogram by height in square meters. This is calculated at 3,6 and 12 month intervals and BMI is calculated at each point of time. Improvement in BMI when compared to the pre-operative BMI is calculated for both the groups and analysed.

SECONDARY OUTCOMES:
Improvement in Type 2 diabetes | 3, 6 and 12 months
  HbA1c for Type 2 diabetes
Improvement in Hypertension | 3, 6, 12 months
  Blood pressure measurement for Hypertension
Improvement in dyslipidemia | 3, 6, 12 months
  Lipid profiles for dyslipidemia
Nutritional status | 3, 6 and 12 months
  Assessed with the skeletal muscle mass
Quality of life of patient | 3, 6 and 12 months
  SF (Short Form) 36 questionnaire
Surgical complications | 3, 6 and 12 months
  Includes postoperative bleeding, 30 day readmission, Leaks, Re-exploration

CONTACTS AND LOCATIONS:
Locations (1):
- GEM Hospital and Research Center, Coimbatore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No